CLINICAL TRIAL: NCT00465595
Title: Psychopharmacology of Psilocybin in Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Heffter Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NA_00001390; Johns Hopkins IRB5 NA_00001390; NCT00850967 (obsolete NCT alias)
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Results first posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-06

CONDITIONS: Depressive Symptoms; Anxiety; Cancer
MeSH Terms: conditions — Depression; Anxiety Disorders; Neoplasms | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Dose First, High Dose Second (Experimental): The Low-Dose-1st Group received the low dose of psilocybin on the first session and the high dose on the second session
  Interventions: Drug: psilocybin
- High Dose First, Low Dose Second (Experimental): The High-Dose-1st Group received the high dose of psilocybin on the first session and the low dose on the second session
  Interventions: Drug: psilocybin

INTERVENTIONS:
Drug: psilocybin — The dose of psilocybin received in the two sessions will range anywhere from low to high.
  Other Names: O-phosphoryl-4-hydroxy-N,N-dimethyltryptamine

SUMMARY:
This research is being done to study the psychological effects of psilocybin in cancer patients. Psilocybin is a naturally occurring substance found in some mushrooms that some cultures have used for centuries in religious practices.

DETAILED DESCRIPTION:
This research is being done to study the psychological effects of psilocybin in cancer patients. Psilocybin is a naturally occurring substance found in some mushrooms that some cultures have used for centuries in religious practices. Psilocybin has not been approved for general medical use by the U.S. Food and Drug Administration (FDA). Its use in this study is investigational. Psilocybin is a mood-altering drug with effects similar to other hallucinogens like LSD and mescaline. Mescaline is the main psychoactive component of the peyote cactus used in Native American religious practices. Such substances have been used for centuries in some cultures as a way of inducing non-ordinary states of consciousness for religious and spiritual purposes.

An earlier study that was done in our lab with healthy participants found that psilocybin, given in a comfortable and supportive setting, can provide an experience that is personally and spiritually meaningful for the participant. This study is being done to find out if psilocybin can also produce personally and spiritually meaningful experiences in cancer patients. This could be important because spirituality has been associated with increased psychological coping and decreased depression in serious illness. People with a diagnosis of cancer between the ages of 21 and 80 years old and who meet the medical requirements may join. About 44 people are expected to take part in this study.

ELIGIBILITY:
Inclusion criteria

Volunteers must:

* Have given written informed consent
* Have a high school level of education
* Be 21 to 80 years old
* Has or has had a cancer diagnosis that is potentially life-threatening. Patients with an active cancer (e.g. stage III or IV with a poor prognosis) or disease progression or recurrence are eligible. Patients who do not have an active cancer or disease progression or disease recurrence are only eligible if at least 1 year has elapsed since their diagnosis.
* Have an ECOG performance status of 0, 1, or 2.
* Have a DSM-IV psychiatric diagnosis, as determined by the SCID, of one or more of the following Axis I psychiatric disorders that is either precipitated by or exacerbated by the psychological stress of the cancer diagnosis: Generalized Anxiety Disorder; Acute Stress Disorder; Post traumatic Stress Disorder; Major Depressive Disorder (mild or moderate severity); Dysthymic Disorder; Adjustment Disorder with Anxiety; Adjustment Disorder with Depressed Mood; Adjustment Disorder with Mixed Anxiety and Depressed Mood; Adjustment Disorder with Disturbance of Conduct; Adjustment Disorder with Disturbance of Emotions and Conduct. Psychiatric diagnosis will be determined by BPRU staff.
* Patients receiving chemotherapy, hormonal therapy, radiation therapy, biologic therapies may participate while receiving those therapies. Continuing hormonal therapy, chemotherapy, or radiation treatment is acceptable if the patient is tolerating the therapy or treatment in a sufficient fashion to allow administration of oral psilocybin.
* Agree that for one week preceding each psilocybin session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the research team. Exceptions will be evaluated by the research team and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.
* Agree not to use nicotine for at least 2 hours before psilocybin administration, and not again until questionnaires have been completed approximately 7 hours after psilocybin administration.
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of psilocybin session days. If the patient does not routinely consume caffeinated beverages, he or she must agree not to do so on psilocybin session days.
* Agree not to take any PRN medications on the mornings of psilocybin sessions, with the exception of daily opioid pain medication. Non-routine PRN medications for treating breakthrough pain that were taken in the 24 hours before the psilocybin session may result in rescheduling the treatment session, with the decision at the discretion of the investigators.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages, within 24 hours of each psilocybin administration. As described elsewhere, exceptions include daily use of caffeine, nicotine, and opioid pain medication.

Exclusion criteria

General Medical Exclusion Criteria

* Cancer with known CNS involvement, or other major CNS disease. In addition to diagnostic results provided by the referring physician, patients will undergo a neurological exam performed by our BPRU internist. Any patient with evidence of a focal deficit will be excluded.
* Hepatic dysfunction as indicated by the following values:

  * GGT > 3 x ULN (upper limit of norm)
  * AST > 3 x ULN
  * ALT > 3 x ULN
  * Tot Bili > 3.0 mg/dl
* Known paraneoplastic syndrome or "ectopic" hormone production by the primary tumor such as the patient could have or be at risk for hypercalcemia, Cushing's syndrome, hypoglycemia, syndrome of inappropriate antidiuretic hormone secretion, or carcinoid syndrome
* Cardiovascular conditions: uncontrolled hypertension, angina, a clinically significant ECG abnormality (e.g. atrial fibrillation), TIA in the last 6 months, stroke, peripheral or pulmonary vascular disease (no active claudication)
* Blood pressure exceeding screening criteria described below
* Epilepsy with history of seizures
* Renal disease (creatinine clearance < 40 ml/min using the Cockcroft and Gault equation)
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Females who are pregnant (positive pregnancy test) or nursing, or are not practicing an effective means of birth control
* Currently taking on a regular (e.g., daily) basis: investigational agents, psychoactive prescription medications (e.g., benzodiazepines), medications having a primary pharmacological effect on serotonin neurons (e.g., ondansetron), or medications that are MAO inhibitors. Long-acting opioid pain medications (e.g. oxycodone sustained release, morphine sustained release -- which are usually taken at 12 hour intervals) will be allowed if the last dose occurred at least 6 hours before psilocybin administration; such medication will not be taken again until at least 6 hours after psilocybin administration.
* For individuals who have intermittent or PRN use of investigational agents, psychoactive prescription medications, medications having a primary pharmacological effect on serotonin neurons, or medications that are MAO inhibitors, psilocybin sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
* In addition to the foregoing, patients will be excluded if they are currently using any the following of potent metabolic inducers or inhibitors: Inducers - Rifamycin (rifampin, rifabutin, rifapentine), anticonvulsants (carbamazepine, phenytoin, Phenobarbital), Nevirapine, Efavirenz, Taxol, Dexamethasone), St Johns Wort; Inhibitors - all HIV protease inhibitors, itraconazole, ketoconazole, erythromycin, clarithromycin, troleandomycin.
* In addition to the foregoing, patients will be excluded if it is a medical requirement that they receive any of the following drugs with low therapeutic index within 12 hours after receiving psilocybin: ergot alkaloids, pimozide, midazolam, triazolam, lovastatin, simvastatin, fentanyl.

Psychiatric Exclusion Criteria

* Individuals with severity of depression or anxiety symptoms warranting immediate treatment with antidepressant or daily anxiolytic medication (e.g., due to suicidal ideation). We will interview patients to determine if referral (e.g., to Community Psychiatry) is necessary. For all individuals who are consented and screened, we will notify the referring physician as to: 1) whether the individual enrolled in the study or not, and 2) if disqualified, why the individual was disqualified. If disqualification was based on severe depression or anxiety (e.g., suicidal ideation), this will be included in the information conveyed to the referring physician. Permission for this contact will be obtained from the participant.
* Current or past history of meeting DSM-IV criteria for Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I or II Disorder
* Current or past history within the last 5 year of meeting DSM-IV criteria for alcohol or drug dependence (excluding caffeine and nicotine).
* Have a first or second degree relative with schizophrenia, psychotic disorder (unless substance induced or due to a medical condition), or bipolar I or II disorder.
* Currently meets DSM-IV criteria for Dissociative Disorder, Anorexia Nervosa, Bulimia Nervosa, or other psychiatric conditions judged to be incompatible with establishment of rapport or safe exposure to psilocybin.

Cardiovascular screening:

There will be at least four blood pressure assessment occasions over at least two separate days. Within a day, assessment occasions will be separated by at least 15 minutes. Each assessment occasion will involve two or more blood pressure readings. To qualify for the study, the mean blood pressure (mm Hg) of the four or more assessment occasions will not exceed 140 systolic and 90 diastolic.

Blood pressure will be taken while subjects are at rest and have been seated or supine for at least 5 minutes. As recommended by the Joint National Committee on Prevention, Detection, Evaluation and Treatment of High Blood Pressure, these assessments will involve the average of 2 or more readings separated by two minutes. If the first 2 readings differ by more than 5 mm Hg, additional readings will be obtained and averaged. On one or more of the blood pressure measurement occasions, the volunteer will be acclimated to the automated blood pressure monitoring equipment by repeatedly taking blood pressure (at least 3 readings) with the device. Because it has been our experience that time-to-time blood pressure readings with the automated equipment can be variable due to measurement artifact, any reading that initially exceeds our threshold value will be reassessed twice within 4 minutes to assure accuracy.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-04; Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland R Griffiths, Ph.D., Principal Investigator — Johns Hopkins School of Medicine, Psychiatry Dept.
Locations (1):
- Behavioral Pharmacology Research Unit, Johns Hopkins Bayview Campus, Baltimore, Maryland, United States

REFERENCES:
- [Result] Griffiths RR, Johnson MW, Carducci MA, Umbricht A, Richards WA, Richards BD, Cosimano MP, Klinedinst MA. Psilocybin produces substantial and sustained decreases in depression and anxiety in patients with life-threatening cancer: A randomized double-blind trial. J Psychopharmacol. 2016 Dec;30(12):1181-1197. doi: 10.1177/0269881116675513. PMID 27909165

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through flyers, internet, and physician referral.
Groups:
- Low-Dose First: The Low-Dose-1st Group received the low dose of psilocybin on the first session and the high dose on the second session.
- High-Dose First: The High-Dose-1st Group received the high dose on the first session and the low dose on the second session.
Period: Overall Study
Arm/Group | Low-Dose First | High-Dose First
Started | 27 | 29
Completed | 22 | 24
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Dose First | High-Dose First | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (11.5) | 56.5 (9.18) | 56.3 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 13 | 13 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 23 | 25 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Education [Count of Participants; unit: Participants]
  High School | 1 | 0 | 1
  College | 8 | 15 | 23
  Post-graduate | 16 | 11 | 27

OUTCOME MEASURES:

1. Primary Outcome: GRID-HAM-D-17 -- Structured Interview Guide for the Hamilton Depression Scale.
Description: The GRID-Hamilton Depression Rating Scale is a 17-item clinician-administered rating scale designed to assess severity of depressive symptoms. The score range for the GRID-HAMD is 0 to 52, with higher score indicating more severe depression. For this clinician-rated measure, a clinically significant response was defined as ⩾50% decrease in measure relative to Baseline; symptom remission was defined as ⩾50% decrease in measure relative to Baseline and a score of ⩽7 on the GRID-HAMD
Time Frame: Baseline, 5 weeks post session 1 and 2, 6-month follow-up
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Low-Dose First Baseline; Low-Dose First Post Session 1; Low-Dose First Post Session 2; Low-Dose First 6 Month: The Low-Dose-1st Group received the low dose of psilocybin on the first session and the high dose on the second session.
- High-Dose First Baseline; High-Dose First Post Session 1; High-Dose First Post Session 2; High-Dose First 6 Month: The High-Dose-1st Group received the high dose on the first session and the low dose on the second session.
Arm/Group | Low-Dose First Baseline | Low-Dose First Post Session 1 | Low-Dose First Post Session 2 | Low-Dose First 6 Month | High-Dose First Baseline | High-Dose First Post Session 1 | High-Dose First Post Session 2 | High-Dose First 6 Month
Number analyzed (Participants) | 25 | 25 | 24 | 22 | 26 | 25 | 25 | 24
units on a scale | 22.32 (.88) | 14.8 (1.45) | 6.5 (.86) | 6.95 (1.24) | 22.84 (.97) | 6.64 (1.04) | 6.52 (1.44) | 6.23 (1.3)

2. Primary Outcome: HAM-A Assessed With the SIGH-A -- a Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A).
Description: The Hamilton Anxiety Rating Scale is a 14-item clinician-administered rating scale designed to assess severity of anxiety symptoms. The score range for the HAM-A is 0 to 56, with higher score indicating more severe anxiety.
  For this clinician-rated measure, a clinically significant response was defined as ⩾50% decrease in measure relative to Baseline; symptom remission was defined as ⩾50% decrease in measure relative to Baseline and a score of ⩽7 on the GRID-HAM-A
Time Frame: Baseline, 5 weeks post session 1 and 2, 6-month follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Low-Dose First Baseline | Low-Dose First Post Session 1 | Low-Dose First Post Session 2 | Low-Dose First 6 Month | High-Dose First Baseline | High-Dose First Post Session 1 | High-Dose First Post Session 2 | High-Dose First 6 Month
Number analyzed (Participants) | 25 | 25 | 24 | 22 | 26 | 25 | 25 | 24
units on a scale | 25.68 (.89) | 16.64 (1.53) | 8.92 (1.14) | 7.95 (1.19) | 25.73 (1.11) | 8.48 (1.16) | 7.52 (1.27) | 7.04 (1.17)

ADVERSE EVENTS:
Groups:
- Low Dose Condition (Group): The experimental design of this study is a complete cross-over, with two groups of participants receiving the low and high doses of psilocybin in counterbalance order. The Low Dose Group is comprised of all low dose psilocybin sessions (n=50). The number of sessions is different from the total enrollment because of dropouts.
- High Dose Condition (Group): The experimental design of this study is a complete cross-over, with two groups of participants receiving the low and high doses of psilocybin in counterbalance order. The High Dose Group is comprised of all high dose psilocybin sessions (n=50). The number of sessions is different from the total enrollment because of dropouts.
Arm/Group | Low Dose Condition (Group) | High Dose Condition (Group)
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 10/56 | 23/56
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Condition (Group) (N=56) | High Dose Condition (Group) (N=56)
Elevated Systolic Blood Pressure (Cardiac disorders) | 9 | 16 — systolic blood pressure higher than 160 at session timepoint
Elevated Diastolic Blood Pressure (Cardiac disorders) | 1 | 7 — Diastolic blood pressure higher than 100 at session timepoint.
Nausea (General disorders) | 0 | 7
Anxiety Episode (Psychiatric disorders) | 7 | 13 — episode isolated to session

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No